CLINICAL TRIAL: NCT02796248
Title: STigma and Its Impact on Glucose Control aMong Youth With diAbetes, a Canada-Wide Study
Acronym: STIGMA
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Kaberi Dasgupta, MD, MSc, FRCP (C), Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: ST-1-16-5046-DK
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes; Social Stigma
Keywords: type 1 diabetes; glucose control; stigma; youth
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Social Stigma | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cross-sectional survey — This is an observation study. Participants will complete a survey at one occasion. Participants are also invited to do a A1c mail-in capillary test.

SUMMARY:
Stigma related to chronic disease is rejection or judgement or exclusion by others that is related to the chronic disease itself and is unwarranted. We are trying to figure out what proportion of young people with type 1 diabetes experience stigma in Canada. By young people, we mean teenagers and young adults; specifically, people who are between 14 and 25 years of age. This is a challenging period in life when identities are developed and peer opinions are felt to be particularly important. Experiencing stigma in this life period may be especially hurtful and may have bad effects on taking care of type 1 diabetes. This may lead to important medical problems like dangerously low or high blood sugar values. By understanding how common stigma is, we can figure out the need for programs and strategies to deal with it.

We will ask young people with type 1 diabetes to help us study this problem by completing an online survey. We will 'advertise' our study through type 1 diabetes clinics, websites, and social media. People who are eligible and interested will click on an internet link and be directed to the survey. Staff at clinics in Montreal, Calgary, and Vancouver will also draw their attention to the posters and/or provide small flyers with the internet link for the study.

Participants will be asked about their general sense of well-being, their habits and behaviours, and their blood sugar control, including frequency of both lows and highs. They will also be asked if they are willing to mail in a small blood sample. If yes, they will receive a kit with a small lancing device and instructions on how to clean their finger tip, prick it, and express a few drops of blood into a small container. They will then mail this back to us in a postage-paid envelope. We will use this to measure their hemoglobin A1c, an overall measure of blood sugar control.

We will use this information to (1) calculate the proportion of young people with type 1 diabetes who experience stigma; (2) figure out what factors and behaviours might predict or signal the experience of stigma; (3) see if there is a link between stigma and A1c control and/or frequent lows by report; (4) explore challenges and solutions voiced through the open-ended questions.

DETAILED DESCRIPTION:
Stigma in diabetes has been understudied. Some recent investigations have examined stigma in adults with type 1 diabetes through in-depth interviews. Such qualitative evaluations provide important insights into the roots and experiences of stigma, but cannot capture the prevalence of the problem. This is a key gap that we will address through a national sample. We will also assess the relationship of stigma to both glycemic control and patient-reported outcomes (PROs) such as mood, self-efficacy, and sense of well-being. PROs are increasingly recognized as critical outcome measures. Finally, we will explore potential solutions with participants.

Methods

1. Selection of questions to capture stigma: As a starting point, we will consider the questions included by Mulvaney and colleagues in their validated Barriers to diabetes adherence in adolescents questionnaire. This 21-item tool includes 6 questions on stigma and 4 other components (stress and burnout, time pressure and planning, social support, parental autonomy support) and showed good overall internal consistency (Cronbach's alpha 0.88). We will also consider additional questions proposed by our team, related to lived experiences with type 1 diabetes and to managing young people with type 1 diabetes (e.g., stigma within social media networks).
2. Creation of on-line questionnaire Based on (1), we will create an online questionnaire through FluidSurveys™ (www.fluidsurveys.com). Participants will be able to fill the survey directly online or offline on tablets, laptops or cell phones. The survey platform also allows participants to upload documents (pictures, videos, text). The questionnaires will be available in both French and English and will include close-ended and open-ended questions. Participants will be allowed to interrupt survey completion as needed and continue at a later time, as convenient.

   In addition to stigma, we will query peer support, quality of life and well-being, diabetes history and current treatment, and socio-demographic information.Overall well-being will be assessed with the WHO-5 well being index, a validated 5-item questionnaire. It is the most widely used questionnaires assessing subjective psychological well-being and has been used in people with type 1 diabetes. Demographic factors including age, sex, and ethnocultural background will be queried to ascertain if the prevalence of diabetes-related stigma is more common in some demographic subgroups (e.g., teens vs. young adults, females vs. males, ethnocultural groups). Similarly, we will query sexual orientation/gender identification in order to ascertain, for example, if being LGBT (i.e., Lesbian, Gay, Bisexual, Transgender), or subgroups thereof, is associated with higher prevalence of diabetes-related stigma. Owing to their potentially sensitive nature, however, the questions on sexual orientation/gender orientation will be explicitly optional

   Following completion of close-ended questions, participants will respond to open-ended questions that seek to capture experiences and perceptions of stigma as well ideas as to how stigma may be effectively addressed. They will be permitted to upload explanatory materials (e.g., videos, testimonials, pictures, drawings).
3. Following survey completion, participants will receive a kit for A1c testing (DTILaboratories, Inc.) with a pre-paid envelope for mailing the sample back to Montreal. The kit includes a sample vial that contains EDTA preservative, a vial holder, a single use lancet, a capillary tube device to draw up a small amount of blood after lancing, and a Ziploc bag. Participants will receive instructions to place the vial on the vial holder, wash their hands, lance a finger tip (they are familiar with this, as type 1 diabetes patients), draw up the blood with the capillary tube, and then release the blood into the vial. The instructions include pictures. They will then place the vial into the Ziploc bag, then into the prelabelled and postage paid box, and then mail the package through a Canada Post mail box. The samples are stable for 2.5 months without refrigeration. The AccuBase A1c Test Kit is a non-fasting, finger stick, whole blood mail-in test requiring a very small blood volume (0.001ml). Samples are stable for 45 days un-refrigerated once collected. They are analysed using a two step process. The screening step detects hemoglobin variants and/or disturbed erythrocyte kinetics by ion-exchange high performance liquid chromatography (HPLC). The second step includes the use of an interference-free procedure HPLC-boronate affinity, that provides a hemoglobin A1c value free of possible interferences including chemically modified derivatives. It is considered one of the most accurate and comprehensive A1c tests available.

Recruitment Adolescents and emerging adults with type 1 diabetes aged ≥ 14 and < 25 years will be recruited. The study will be publicized through Facebook©, Twitter© , and other forms of social media as well as websites of organizations such as Canadian Diabetes Association, Juvenil Diabetes Research Foundation, Diabète Québec and the Quebec Diabetic Children's Foundation. These organizations may be asked to mail out flyers or send email messages through any patient contacts. Specifically, the study will be publicized through posters at diabetes clinics, Facebook© pages and websites of diabetes organizations and messages on Twitter©. As in previous studies, we will include a description of the STIGMA study with a link on the websites of diabetes organizations. We will also ask the organizations to contact their members directly to inform them about the study, with a link embedded in the email message.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* Canadian citizen
* Aged between 14 and 24 years

Exclusion Criteria:

* other forms of diabetes

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults (14-24 years of age) with type 1 diabetes living in Canada
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Presence of stigma | At survey completion
  Will be ascertained through a series of questions

SECONDARY OUTCOMES:
A1c | At survey completion
  As noted, participants will be provided with a lancet and small container in which to express a couple of drops of blood. While this may cause some discomfort, given that all participants have type 1 diabetes, they are familiar with this procedure and express blood in this fashion regularly.
Hypoglycemia frequency | At survey completion; recall period varies from past week to past year
  Questions
Diabetes-related self-efficicay | At survey completion
  Questions based on Iannotti et al,. Developmental and Behavioral Pediatrics, 2006
Diabetes-related distress | At survey completion
  Questions based on Polonsky et al, Diabetes Care, 1995
Quality of life | At survey completion; recall period is past month
  Questions based on Varni et al. Diabetes Care 2003
Well-Being Index | At survey completion; recall period is past two months
  Questions from World Health Organization WHO (Five) Well-Being Index

CONTACTS AND LOCATIONS:
Overall Officials: Kaberi Dasgupta, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (4):
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brazeau AS, Nakhla M, Wright M, Henderson M, Panagiotopoulos C, Pacaud D, Kearns P, Rahme E, Da Costa D, Dasgupta K. Stigma and Its Association With Glycemic Control and Hypoglycemia in Adolescents and Young Adults With Type 1 Diabetes: Cross-Sectional Study. J Med Internet Res. 2018 Apr 20;20(4):e151. doi: 10.2196/jmir.9432. PMID 29678801
- [Background] Brazeau AS, Nakhla M, Wright M, Panagiotopoulos C, Pacaud D, Henderson M, Rahme E, Da Costa D, Dasgupta K. Stigma and Its Impact on Glucose Control Among Youth With Diabetes: Protocol for a Canada-Wide Study. JMIR Res Protoc. 2016 Dec 15;5(4):e242. doi: 10.2196/resprot.6629. PMID 27979791